CLINICAL TRIAL: NCT02291796
Title: Early Effect Of Bezafibrate On Fibrinogen Levels, Inflammatory Response And Clinical Impact, In Patients With ST Elevation Acute Myocardial Infarction
Brief Title: Bezafibrate for Hyperfibrinogenemia in Acute Myocardial Infarction
Acronym: BEZAFIBRAMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Maria Alejandra Madrid Miller, Head of the Division of Health Research, UMAE Hospital de Cardiologia, Centro Médico Nacional Siglo XXI, IMSS, México, D.F., Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2010-3604-17
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Bezafibrate; Hyperfibrinogenemia; Inflammatory response; Acute myocardial infarction; Mayor cardiovascular events
MeSH Terms: interventions — Bezafibrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bezafibrate group (Experimental): Patients with acute coronary syndrome with ST elevation and fibrinogen receiving a dose of 400 mg every 24 hours of Bezafibrate in addition to conventional anti-ischemic treatment
  Interventions: Drug: Bezafibrate
- Control group (No Intervention): Patients with acute coronary syndrome with ST elevation and hyperfibrinogenemia who received only conventional anti-ischemic treatment

INTERVENTIONS:
Drug: Bezafibrate — Patients with ST elevation acute myocardial infarction (STEAMI) and with fibrinogen concentration >500 mg/dl at 72 h of evolution, were randomly assigned to bezafibrate 400 mg/day or just conventional therapy
  Arms: Bezafibrate group

SUMMARY:
Introduction: Plasma fibrinogen levels have been identified as an important risk factor for cardiovascular diseases and could have a prognostic value. Bezafibrate decreases fibrinogen levels and also the incidence of major cardiovascular events in primary prevention, but its effects in acute coronary syndrome is unknown.

Hypothesis: Bezafibrate effect over statin therapy reduces fibrinogen concentrations, inflammatory response and clinical events, in patients with ST segment elevation ACS and hyperfibrinogenemia.

Methods: In a randomized clinical trial, controlled with conventional therapy. Patients with ST elevation acute myocardial infarction (STEAMI) and with fibrinogen concentration >500 mg/dl at 72 h of evolution, were randomly assigned to bezafibrate 400 mg/day (group I n=50) or just conventional therapy (group II n=50). Serum fibrinogen, c reactive protein and cytokines were measured. Clinical end points were recurrence of angina or infarction, left ventricular failure, cardiovascular mortality and combined end points during hospitalization.

DETAILED DESCRIPTION:
Patients >18 years of age who were admitted to the Cardiovascular Intensive Care Unit of the Cardiology Hospital, National Medical Center, Century XXI (Mexico City) and diagnosed with ST segment elevation Acute Coronary Syndrome (ACS) and hyperfibrinogenemia within 72 h of symptom onset were included. Acute myocardial infarction (AMI) was diagnosed when high myocardial necrosis markers were found such as CPK total >150% basal value or troponin I ≥1 ng/ml plus one of the following: ischemic precordial pain >30 min with/without dyspnea, diaphoresis, nausea, vomiting, or ST segment elevation >1 mm in two or more contiguous leads or left bundle branch block, new or presumed new. Hyperfibrinogenemia was diagnosed after fibrinogen concentrations reached >500 mg/dl at 72 h of evolution. All patients signed an informed consent form to participate in the study.

Patients with known bezafibrate allergy, previous fibrate treatments, patients with cardiogenic shock, hepatic failure, renal failure, history of neoplastic disease, chronic inflammatory disease or active infectious process, anti-inflammatory or immunosuppressive therapies, fibrinolysis with streptokinase and patients with triglyceride concentrations >150 mg/dl were excluded.

Patients were classified into two groups: group I, patients who received a 400-mg bezafibrate dose every 24 h plus conventional anti-ischemic therapy; and group II, patients who only received conventional anti-ischemic therapy. Patients were assigned to each group using random numbers tables. Conventional adjunctive anti-ischemic therapy included dual antiplatelet therapy, antithrombotic, beta blockers, statins, angiotensin converting enzyme inhibitors, and others according to each case. Twelve-lead ECG was carried out daily and under recurrent ischemic event. Laboratory tests were also carried out including cardiac enzymes, lipid profile and CRP.

Our goal was to determine if bezafibrate therapy combined with conventional anti-ischemic therapy reduces fibrinogen levels. Primary endpoints were recurrent ischemic event such as reinfarction or post-infarction angina and left ventricular failure. Secondary endpoints were death, need for revascularization and combined clinical endpoints that will be presented after randomization and before patient discharge.

Blood samples were taken in all patients by venipuncture in an upper extremity (Vena basilica, cephalic or any tax): 4.5 ml of blood, collected into a 0.5 ml tube vacutainer with sodium citrate buffer (9: 1) 0129 M 3.8% (blue top), which is used to determine the coagulation time and fibrinogen; and another 7 ml, which will be collected in vacutainer tubes dry (red cap). The samples will be centrifuged at 2000 rpm for 10 min and the serum obtained will be divided into aliquots of 200 ul to keep at -70 ° C for subsequent biochemical determinations. This procedure will be performed on admission to the Cardiovascular Intensive Care Unit and on days 5, 7 and 30 of its randomizationAll patients after hospital discharge, will be cited by telephone at 30 days after randomization, for taking blood samples, as well as for clinical evaluation.Fibrinogen Determination All venous blood samples (4.5 ml) will be taken from an upper limb (basilic vein, cephalic vein or any of their tributaries) and collected in a Vacutainer (Becton Dickinson, Franklin Lakes, NJ) tube with 0.5 ml sodium nitrate buffer (9:1) 0.129 M 3.8% (blue top). This procedure was repeated at discharge or after 7 days when the patient was subjected to a long hospital stay. PT-Fibrinogen HS Plus kit (Beckman Coulter, Brea, CA) was used. This contains high-sensitivity calcium thromboplastin to determine prothrombin time and fibrinogen and to evaluate extrinsic pathway of coagulation in citrated human plasma using an auto-analyzer ACL-800 (Cobas, Roche Diagnostics, Indianapolis, IN) where fibrinogen levels are determined through turbidimetry. Test measure correlation was r = 0.95. Units reported for fibrinogen are mg/dl and the standard control is 273 mg/dl with a linearity of 700 mg/dl.

c) Clinical evaluation For clinical follow-up evaluation after randomization, the presence of recurrent cardiovascular events and is regarded as secondary endpoints: events of recurrent ischemia either the presence of angina, reinfarction, or silent ischemia, need for procedures Emergency myocardial revascularization left ventricular failure, shock and death, stating the time from randomization to the presentation of the event, electrocardiographic or biochemical changes that occur time. Both during their hospital stay, as at discharge, data were obtained either directly by history, physical examination and laboratory, and the clinical record, taking into account the assessment of the treating physician and recorded in the data collection sheet.

Cytokines assay Concentration of cytokines (IL-8, IL-1β, IL-6, IL-10, TNF e IL-12) were measured by ELISA system (Biosource), with two different monoclonal antibodies against different epitopes of interleukins, biotinylated detector antibodies, conjugated Streptavidin-HRP (SAV) buffer, chromogen substrate and stop solution. Once the plasma samples and the supernatants were unfroze, all the standard and samples were diluted with the standard dilutor assay buffer. A100μl of the standard, samples, supernatants and controls were added to a coated microtiter plate by duplicate test and incubated by an hour. The biotinylated detector antibodies were diluted in buffer and added 50μl to 100 μl to each well, excepted the empty chromogen, then incubated for 1 hour at 37°C. Plates were the washed; a 100 μl of SAV diluted with buffer, was added to each well and incubated for other 45 min. Microtiter plate was washed again. Tetramethylbenzidine substrate was added (100 μl each well), incubated for 15min more in darkness at room temperature. Finally 50 to 100 μl of stop solution was used. Plates were read 30 min after, at 490 nm in an automated microplate reader.

Statistical Analysis Continuous variables were described according to distribution (mean ± standard deviation, median and percentiles). Demographic characteristics of the population were expressed in frequency percentage. Student t-distribution was used for bivariate analysis of continuous variables and group comparison for those parameters with normal distribution and Mann-Whitney U test for those with non-normal distribution. Wilcoxon test was used to analyze the fibrinogen concentration difference within each group. Dichotomous variables were tested using X2 and Fisher's exact test depending on expected values. Relative risk (RR) and 95% confidence intervals (CI) were calculated. Multivariate analysis adjusted for potential confounders will be performed. Calculation of the number needed to treat and the analysis with intention to treat will be done. Relative risks and confidence interval of 95% will be calculated. The value p, equal or less to 0.05, will be consider significant. SPSS v.20.0 software will be used for data analysis

Ethical considerations The study will be evaluated by the Research Committee and Local Research Ethics in Health UMAE Cardiology Hospital National Medical Center Siglo XXI, for approval. The study conforms to the standards set by the Declaration of Helsinki, the rules of the General Health Law in research in our country and the Good Clinical Practice of the International Conference on Harmonization.

The study considered more than minimal risk and its main objective is to evaluate the additive effect of bezafibrate to conventional anti-ischemic drug therapy in patients with acute coronary syndrome with ST segment elevation.

Bezafibrate is a drug that is in the institutional basic list, is used to provide treatment for patients with dyslipidemia, particularly in patients with hypertriglyceridemia. During the study, there were not changes or interventions against the standard treatment prescribed by the treating physician, which has proven benefits according to the Clinical Practice Guidelines for the treatment of patients with acute coronary syndrome with ST segment elevation.

In accordance with the provisions of the Belmont Report, can be carried out in conjunction with the usual therapeutic practices used in these patients, since it is designed to assess the safety and efficacy of a therapy, however it will be subject to formal investigation in order to determine its safety and effectiveness for protection of those involved.

Adverse events reported in general are rare, transient and mild to moderate intensity. The adverse reactions reported most frequently are loss of appetite (about 1.8%); with less frequency (1 case in 1,000 patients who take the bezafibrate) abdominal pain, nausea diarrhea, distension of the stomach, erectile dysfunction, feeling dizzy, gastrointestinal problems, hair loss, headaches, abnormal laboratory test results, anaphylactic reactions, hypersensitivity reactions, itching, kidney problems, muscle problems including muscle weakness, cramps, pain or tenderness, photosensitivity skin reaction, skin rash or rashes, urticaria. Other uncommon side effects (more than 1 in 10,000 people who take bezafibrate) are neuropathy of the extremities, pancreatitis, paraesthesiae. dizziness,. There are reported very rare, fewer than 1 in 10,000 patients receiving bezafibrate, of blood problems, erythema multiforme, gallstones, lung problems, rhabdomyolysis, Stevens-Johnson syndrome, toxic epidermal necrolysis, unexplained or easy bruising of the skin or mucous membranes.

During the study, patients in addition to conventional studies of 12-lead electrocardiogram at rest, echocardiography, X-rays and laboratory tests, need the venous blood samples for serial measurements of fibrinogen, C-reactive protein and serum proinflammatory cytokines, at 5, 7 and 30 days after randomization.

Patients who meet the selection criteria will be included. No patients were included in critical condition or hemodynamic decompensation. All patients were requested to sign for informed consent after explaining potential risks and benefits of treatment. They were explained in detail, what it will be patient participation in the study, assessment processes and monitoring to be performed, as well as the actions to be carried out in case of any adverse events. The invitation to participate and signed consent application will be requested by a different doctor than the treating physician. It will make the clarification to the patient that their participation in the study is completely voluntary and if so manifest, may withdraw from the study at any time If the patient has an adverse drug event may be addressed immediately in the emergency department of the Hospital UMAE Cardiology. The corresponding report of any side effects will to be performed to the committee of pharmaco-vigilance (hospital committee), the VENCER system (Institutional system for reports of any adverse event, side effect and pharmacology interaction) ant to the COFEPRIS (that is the national Committee). The side effects are part of the study analysis for the evaluation of drug safety. The patient shall record in a log any side or adverse event occurring during the treatment time and given a telephone number to contact the physician 24 hours a day during the six months being treated with bezafibrate, and time duration of the study. The patient may also contact the physician if any questions regarding the study.

The patient data will be handled confidentially and no personal information that could identify them will be used, in case of distribution and publication of results. Every patient is assigned a serial number according to the time of study entry to identify him in subsequent evaluations.

Because the drug used is part of the basic list of the IMSS, there is no conflicts of interest among researchers.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age who were admitted to the Cardiovascular Intensive Care Unit of the Cardiology Hospital, National Medical Center, Century XXI (Mexico City) and diagnosed with ST segment elevation ACS and hyperfibrinogenemia within 72 h of symptom onset

Exclusion Criteria:

* Patients with known bezafibrate allergy,
* previous fibrate treatments,
* patients with cardiogenic shock,
* hepatic failure,
* renal failure,
* history of neoplastic disease,
* chronic inflammatory disease or active infectious process,
* anti-inflammatory or immunosuppressive therapies,
* fibrinolysis with streptokinase and
* patients with triglyceride concentrations >150 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Fibrinogen levels | From hospital stay to 3 months
  PT-Fibrinogen HS Plus kit (Beckman Coulter, Brea, CA) to determine prothrombin time and fibrinogen and to evaluate extrinsic pathway of coagulation in citrated human plasma using an auto-analyzer ACL-800 (Cobas, Roche Diagnostics, Indianapolis, IN) where fibrinogen levels are determined through turbidimetry.
Inflammatory response | From hospital stay to 1 month
  Concentration of cytokines (IL-8, IL-1β, IL-6, IL-10, TNF e IL-12) measured by ELISA system (Biosource)

SECONDARY OUTCOMES:
Recurrence of major cardiovascular events | From hospital stay to 1 month
  angina, reinfarction, heart failure, death, and combined endpoints
Safety of treatment with bezafibrate (Any side effect that comes with the intake of bezafibrate) | From hospital stay to 1 month
  Any side effect that comes with the intake of bezafibrate

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Madrid-Miller, MD, Principal Investigator — Head of the Division of Health Research UMAE Hospital de Cardiologia, Centro Médico Nacional Siglo XXI, IMSS